CLINICAL TRIAL: NCT05352815
Title: A 52 Week Study Comparing the Efficacy and Safety of Once Weekly IcoSema and Once Weekly Insulin Icodec, Both Treatment Arms With or Without Oral Anti Diabetic Drugs, in Participants With Type 2 Diabetes Inadequately Controlled With Daily Basal Insulin.
Brief Title: A Research Study to See How Well the New Weekly Medicine IcoSema, Which is a Combination of Insulin Icodec and Semaglutide, Controls Blood Sugar Level in People With Type 2 Diabetes Compared to Weekly Insulin Icodec
Acronym: COMBINE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1535-4591; U1111-1260-8259 (Other: World Health Organization (WHO)); 2020-005281-34 (EudraCT Number)
Record Dates: First submitted 2022-04-24; First posted 2022-04-29 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IcoSema (Experimental)
  Interventions: Drug: IcoSema
- Insulin icodec (Active Comparator)
  Interventions: Drug: Insulin icodec

INTERVENTIONS:
Drug: IcoSema — Participants will receive once weekly IcoSema subcutanously (s.c. under the skin) with or without oral anti diabetic drugs for 52 weeks.
  Arms: IcoSema
Drug: Insulin icodec — Participants will receive once weekly Insulin icodec subcutanously (s.c. under the skin) with or without oral anti diabetic drugs for 52 weeks.
  Arms: Insulin icodec

SUMMARY:
This study will compare the new medicine IcoSema, which is a combination of insulin icodec and semaglutide, taken once a week, to insulin icodec taken once a week in people with type 2 diabetes.

The study will look at how well IcoSema controls blood sugar level in people with type 2 diabetes compared to insulin icodec.

Participants will either get IcoSema or insulin icodec. Which treatment participants get is decided by chance. IcoSema and insulin icodec are both new medicines that doctors cannot prescribe.

Participants will get IcoSema or insulin icodec, which participants must inject once a week with a pen, which has a small needle, in a skin fold in the thigh, upper arm, or stomach.

The study will last for about 1 year and 1 month. Participants will have 21 clinic visits, 31 phone/video calls with the study doctor, and 4 contacts with the site that can either be clinic visits or phone/video calls At 11 clinic visits participants will have blood samples taken. At 7 clinic visits participants cannot eat or drink (except for water) for 8 hours before the visit.

Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

Not applicable for China: Participants will be asked to wear a sensor that measures their blood sugar level all the time during a 5 week period at the end of the study.

ELIGIBILITY:
Key inclusion criteria

1. Male or female and age above or equal to 18 years at the time of signing informed consent.
2. Diagnosed with type 2 diabetes mellitus 180 days or more before screening.
3. HbA1c of 7.0 10.0% (53.0 85.8 mmol/mol) (both inclusive) as assessed by central laboratory on the day of screening.
4. Treated with once daily or twice daily basal insulin (neutral protamine hagedorn insulin, insulin degludec, insulin detemir, insulin glargine 100 units/mL, or insulin glargine 300 units/mL) 20- 80 units/day for 90 days or more before screening. Short term bolus insulin treatment for a maximum of 14 days before screening is allowed, as is prior insulin treatment for gestational diabetes. The treatment can be with or without any of the following anti diabetic drugs with stable doses for 90 days or more before screening:

   * Metformin
   * Sulfonylureas (a)
   * Meglitinides (glinides) (a)
   * DPP 4 inhibitors (a)
   * Sodium glucose co transporter 2 inhibitors
   * Alpha glucosidase inhibitors
   * Thiazolidinediones
   * Marketed oral combination products only including the products listed above.
5. Body mass index (BMI) below or equal to 40.0 kg/m^2. (a) Sulfonylureas, meglitinides (glinides) and DPP 4 inhibitors must be discontinued at randomisation.

Key exclusion criteria

1. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
2. Anticipated initiation or change in concomitant medication (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or systemic corticosteroids).
3. Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening.
4. Any episodes (as declared by the participant or in the medical records.) of diabetic ketoacidosis within 90 days before screening.
5. Presence or history of pancreatitis (acute or chronic) within 180 days before screening.
6. Any of the following: Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days before screening.
7. Chronic heart failure classified as being in New York Heart Association Class IV at screening.
8. Recurrent severe hypoglycaemic episodes within the last year (12 months) as judged by the investigator.
9. Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days before screening or in the period between screening and randomisation. Pharmacological pupil dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1291 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (280):
- United States (109):
  - Pri Med Grp dba/Gil Ctr Fam, Gilbert, Arizona
  - Lenzmeier Fam Med CCT Research, Glendale, Arizona
  - Phoenician Centers for Research & Innovation PCRI, Phoenix, Arizona
  - Medical Investigations, Inc., Little Rock, Arkansas
  - John Muir Physicians Network, Concord, California
  - Headlands Research California, LLC, Escondido, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Clinical Trials Research_Sacramento, Lincoln, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Downtown LA Res Ctr. Inc., Los Angeles, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Clinical Trials Research_Sacramento_0, Sacramento, California
  - San Diego Family Care, San Diego, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Clinical Res Of W Florida Inc, Clearwater, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - University of Miami, Miami, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Suncoast Clin Res Port Richey, New Port Richey, Florida
  - Clinical Neuroscience Solution, Orlando, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Javara/Privia Med Grp GA,LLC, Albany, Georgia
  - Emory University SOM, Atlanta, Georgia
  - Javara Inc., Fayetteville, Georgia
  - Physicians Research Assoc. LLC, Lawrenceville, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Saltzer Medical Group Research, Nampa, Idaho
  - UnityPoint Health-Diabetes Care Center, Peoria, Illinois
  - Endeavor Health, Skokie, Illinois
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Cotton O'Neil Diab & Endo Ctr, Topeka, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Barnum Medical Research Inc., Natchitoches, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Ileana J Tandron APMC, Slidell, Louisiana
  - MedStar Hlth Res Institute, Hyattsville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - MassResearch, LLC, Waltham, Massachusetts
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - Elite Research Center, Flint, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Jefferson City Medical Group, PC, Jefferson City, Missouri
  - Methodist Phys. Clinic, Omaha, Nebraska
  - University of NE Med Ctr, Omaha, Nebraska
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Palm Research Center Inc., Las Vegas, Nevada
  - Southern New Hampshire Diabete, Nashua, New Hampshire
  - John J Shelmet, MD, Lawrenceville, New Jersey
  - Albuquerque Clin Trials, Inc., Albuquerque, New Mexico
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Javara Inc. / Tryon Medical Partners PLLC, Charlotte, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Central Ohio Clinical Research LLC, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Intend Research, Norman, Oklahoma
  - Care Access, Warwick, Rhode Island
  - Palmetto Clinical Research, Summerville, South Carolina
  - Athens Medical Group, Athens, Tennessee
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - Holston Medical Group_Bristol, Bristol, Tennessee
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - HealthStar Physicians PC, Morristown, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Texas Diabetes & Endocrinology, P.A._Austin, Austin, Texas
  - Osvaldo A. Brusco MD PA, Corpus Christi, Texas
  - Cedar Research, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Univ of TX SW Med Ctr Dallas, Dallas, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Javara Inc. / Privia Medical Group Gulf Coast PLLC, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Medical Colleagues-Texas LLP, Katy, Texas
  - Andres Garcia-Zuniga, MD, P.A, Laredo, Texas
  - Milton Haber, M.D., Laredo, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Clinical Investigations Of Texas, Plano, Texas
  - Texas Diabetes &Endocrinology, Round Rock, Texas
  - Sun Research Institute, San Antonio, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - Diabetes & Gladular Disease Research A Cetero Research Co, San Antonio, Texas
  - Diabetes Glandular Diseases Clinic, San Antonio, Texas
  - Javara Inc Privia Grp Gulf Cst, San Marcos, Texas
  - SimCare, PLLC, Sugar Land, Texas
  - Sugar Lakes Family Practice PA, Sugar Land, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Javara Inc. / Privia Medical Group LLC_Appomattox, Appomattox, Virginia
  - Javara Inc/Privia Md GpLLC Fst, Forest, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Amherst Family Practice P.C., Winchester, Virginia
  - Sound Medical Research, Port Orchard, Washington
  - Rainier Clin Res Ctr Inc, Renton, Washington
  - Ascension Columbia St. Mary's Hospital, Milwaukee, Wisconsin
- Australia (10):
  - The Canberra Hospital_Garran, Garran, Australian Capital Territory
  - Holdsworth House Clinical Research, Darlinghurst, New South Wales
  - Momentum Clinical Research Darlinghurst, Darlinghurst, New South Wales
  - Novatrials, Kotara, New South Wales
  - Illawarra Diabetes Service Clinical Trials & Research Unit, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Barwon Health (The Geelong Hospital), Geelong, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (7):
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - UZ Brussel - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc - Serv Endocrinologie - Diabétologie, Brussels
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - AZ Groeninge - Kortrijk - Centrum Endo - Diabetologie, Kortrijk
  - CHU Tivoli, La Louvière
  - UZ Leuven - Endocrinology, Leuven
- Bulgaria (5):
  - IPSMC - Dr. Nikolay Kostadinov EOOD, Burgas
  - Medical center Medi City 21 OOD, Kyustendil
  - DCC I- Pleven EOOD Endocrinology, Pleven
  - UMHAT Kaspela EOOD, Endocrinology and Metabolic Diseases Clinic, Plovdiv
  - MMA-MHAT Sofia, Clinic of Endocrinology and Metab. Diseases, Sofia
- China (17):
  - Anhui Provincial Hospital-Endocrinology, Hefei, Anhui
  - Peking University People's Hospital-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Huizhou Central People's Hospital-Endocrinology, Huizhou, Guangdong
  - Harrison International Peace Hospital, Hengshui, Hebei
  - Hengshui People's Hospital (Harrison International Peace Hospital)-Endocrinology, Hengshui, Hebei
  - Huaihe Hospital of Henan University-Endocrinology, Kaifeng, Henan
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University_Nanjing, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University-Endocrinology, Suzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shanghai Fifth People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University-Endocrinology, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
- Croatia (5):
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - Poliklinika SLAVONIJA OSIJEK, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Osijek, Osijek
  - Opca bolnica Pula, Pula
  - KBC Rijeka, Endokrinologija, Rijeka
- Finland (6):
  - Ähtärin terveysasema, Ähtäri
  - Health Step Finland Oy, Kuopio
  - Etelä-Savon sosiaali- ja terveyspalvelujen kuntayhtymä, Mikkeli
  - Raision sosiaali- ja terveyskeskus, Raisio
  - Tampereen diabetesvastaanotto, Tampere
  - Turku University Hospital, Turku
- India (23):
  - Yashoda Hospital, Secunderabad, Andhra Pradesh
  - Apollo Excelcare Hospital, Guwahati, Assam
  - Gujarat Endocrine Centre, Ahmedabad, Gujarat
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Lifecare Hospital and Research Centre, Bangalore, Karnataka
  - Mysore Medical College and Research Institute, Mysore, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Jothydev's Diabetes & Research Center, Thriruvananthapuram, Kerala
  - TOTALL Diabetes Hormone Institute, Indore, Madhya Pradesh
  - Excel Endocrine Centre, Kolhāpur, Maharashtra
  - BYL Nair Hospital and T N Medical College Department of endo, Mumbai, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Bhaktivedanta Hospital & Research Institute, Mumbai, Maharashtra
  - Inamdar Multispeciality Hospital, Pune, Maharashtra
  - S.C.B. Medical College, Cuttack, Odisha
  - Post Graduate Institute of Medical Education & Research, Chandigarh, Punjab
  - Dayanand Medical College & Hospital_Ludhiana, Ludhiana, Punjab
  - M.V.Hospital for Diabetes Pvt. Ltd., Chennai, Tamil Nadu
  - Arthur Asirvatham hospital,, Madurai, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - Ramdev Rao Hospital, Hyderabad, Telangana
  - Lady Hardinge Medical College, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
- Italy (6):
  - A.O.U. Consorziale Policlinico di Bari, Bari, BA
  - Pol. Uni. Campus Biomedico, Roma, RM
  - Policlinico Mater Domini Università di Catanzaro, Catanzaro
  - ASL 4 Chiavarese, Chiavari (genova)
  - Ospedale Policlinico San Martino, Genova
  - Grande Ospedale Metropolitano Niguarda, Milan
- Japan (18):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Japan
  - Manda Memorial Hospital_Internal Medicine, Sapporo-shi, Hokkaido, Hokkaido, Japan
  - Hayashi Diabetes Clinic, Chigasaki-shi, Kanagawa, Kanagawa, Japan
  - Hayashi Diabetes Clinic_Internal Medicine and Diabetes Medicine, Chigasaki-shi, Kanagawa, Japan
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - Heiwadai Hospital, Miyazaki, Miyazaki
  - Kumanomae Nishimura Naika Clinic_Internal Medicine, Arakawa-ku, Tokyo
  - Akaicho Clinic, Chiba-shi, Chiba
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Futata Tetsuhiro Clinic Meinohama, Fukuoka-shi, Fukuoka
  - Kunisaki Makoto Clinic, Fukuoka-shi, Fukuoka
  - Sasaki Internal Medicine, Hokkaido
  - Yoshimura clinic, Kumamoto
  - Hisatomi Clinic, Saga-shi, Saga
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Yokohama City University Hospital, Endocrinology, Metabolism, Yokohama-shi, Kanagawa
- Mexico (3):
  - Hospital Universitario Dr. José Eleuterio González_Monterrey, Monterrey, Nuevo León
  - Centro de Investigación Cardiometabólica de Aguascalientes, Aguascalientes
  - Clínicos Asociados BOCM, S.C., Mexico City
- Norway (7):
  - Nordlandssykehuset Bodø, Bodø
  - Drammen sykehus - Vestre Viken HF, Drammen
  - Bærum sykehus, Gjettum
  - Sykehuset Innlandet HF Hamar, Hamar
  - Akershus universitetssykehus HF, Lørenskog
  - Oslo universitetssykehus Aker, Oslo
  - St. Olavs Hospital HF, Trondheim
- Poland (4):
  - NZOZ Przychodnia Specjalistyczna Medica, Lublin, Lubelski
  - Uniwersyteckie Centrum Kliniczne (UCK), Gdansk
  - NZOZ "CenterMed Lublin" Sp. z o.o., Lublin
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
- Portugal (12):
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - Unidade Local De Saude De Almada-Seixal E.P.E. - Hospital Garcia de Orta, Almada
  - Unidade Local De Saude De Amadora Sintra E.P.E. - Hospital Prof. Dr. Fernando da Fonseca, Amadora
  - Unidade Local De Saude Da Regiao De Aveiro E.P.E., Aveiro
  - Unidade de Local de Saúde de Braga, Braga
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital Egas Moniz, Lisbon
  - Hospital Da Luz S.A., Lisbon
  - Unidade Local de Saúde de Matosinhos, Matosinhos Municipality
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Hospital Luz Arrabida, S.A., Vila Nova de Gaia
  - Unidade Local De Saude De Tras-Os-Montes E Alto Douro E.P.E., Vila Real
- Puerto Rico (2):
  - Advanced Clinical Research LLC, Bayamón
  - Manati Ctr For Clin Research, Manatí
- Romania (6):
  - Institutul National De Diabet Nutritie Si Boli Metabolice Prof.Dr.N.Paulescu Bucuresti- Ion Movila, Bucharest, Bucurestii
  - CMI Diabet, Nutritie, Boli Metabolice "Dr Pop Lavinia", Baia Mare, Maramureş
  - Mariodiab Clinic SRL, Brasov
  - SC Consultmed SRL, Iași
  - Clinica Korall S.R.L. Satu Mare, Satu Mare
  - Spitalul Judetean De Urgenta Sfantul Ioan Cel Nou Suceava, Suceava
- Russia (7):
  - Tumen State Medical University, Tyumen, Russia
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - Limited Liability Company "AriVa-Med", Kursk
  - City Consultative & Diagnostic Centre #1, Saint Petersburg
  - Saratov regional clinical hospital, Saratov
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade, Serbia
- South Africa (7):
  - Deepak Lakha, Johannesburg, Gauteng
  - Hemant Makan, Johannesburg, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Dr Pillay's Rooms, Durban, KwaZulu-Natal
  - Armansis Medical Centre, Brits, North West
  - Langeberg Clinical Trials, Cape Town, Western Cape
  - Netcare Alberton Hospital, Alberton
- South Korea (13):
  - Soonchunhyang University Hospital, Cheonan, Chungcheongnam-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital_Seongnam-si, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Taiwan (5):
  - Changhua Christian Hospital_Metabolic Dept., Changhua
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Taipei Medical University Hospital, Taipei
- Turkey (Türkiye) (7):
  - Ankara Üniversitesi Tıp Fakültesi İbni Sina Hastanesi-Endokrinoloji, Ankara, Altindag
  - Çukurova Üniversitesi Tıp Fakültesi Balcalı Hastanesi- Endokrinoloji, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Haseki Eğitim ve Araştırma Hastanesi- Dahiliye, Istanbul
  - Göztepe Prof. Dr.Süleyman Yalçın Şehir Hastanesi- Dahiliye, Istanbul
  - T.C. S.B. Ist Il SagMud Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Tekirdağ Namık Kemal Üniversitesi Hastanesi- Dahiliye, Tekirdağ

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Mathieu C, Giorgino F, Kim SG, Larsen JH, Philis-Tsimikas A, Ramachandran A, Pagliaro Rocha TM, Shankarappa VB, Terauchi Y, Ji L. Once-weekly IcoSema versus once-weekly insulin icodec in type 2 diabetes management (COMBINE 1): an open-label, multicentre, treat-to-target, randomised, phase 3a trial. Lancet Diabetes Endocrinol. 2025 Jul;13(7):568-579. doi: 10.1016/S2213-8587(25)00096-8. Epub 2025 Jun 4. PMID 40482671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 192 sites in 20 countries.
Pre-assignment Details: Participants with type 2 diabetes (T2D) inadequately controlled with daily basal insulin were randomised in 1:1 ratio to receive subcutaneous (s.c.) injection of IcoSema or insulin icodec once weekly with or without oral anti-diabetic drugs (OADs).
Groups:
- IcoSema: Participants received once-weekly subcutaneous injections of 700 units per milliliter (U/mL) of insulin icodec and 2 milligrams per milliliter (mg/mL) of semaglutide for 52 weeks.
- Insulin Icodec: Participants received once-weekly subcutaneous injections of 700 U/mL of insulin icodec for 52 weeks.
Period: Overall Study
Arm/Group | IcoSema | Insulin Icodec
Started | 646 | 645
Treated | 644 | 644
Full Analysis Set | 646 | 645
Safety Analysis Set | 644 | 644
Completed | 611 | 611
Not Completed | 35 | 34
Not completed — Withdrawal by Subject | 28 | 24
Not completed — Lost to Follow-up | 4 | 7
Not completed — Death | 2 | 3
Not completed — Site closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | IcoSema | Insulin Icodec | Total
Number analyzed (Participants) | 646 | 645 | 1291
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (10.5) | 60.7 (10.2) | 60.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 246 | 492
  Male | 400 | 399 | 799
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 101 | 110 | 211
  Not Hispanic or Latino | 545 | 535 | 1080
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 1 | 6
  Asian | 216 | 204 | 420
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 19 | 25 | 44
  White | 404 | 410 | 814
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change from baseline (week 0) to week 52 in HbA1c is presented. The outcome measure was evaluated based on the data from in study period, where all data from randomisation until last date of any of the following: 1) last direct participant-site contact; 2) participants who withdrew their informed consent; 3) last participant-investigator contact as defined by the investigator for participants who lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death of participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 52
Population: Full Analysis Set (FAS) included all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 598 | 605
Percentage point of HbA1c | -1.60 (0.99) | -0.90 (1.01)
Statistical Analysis 1: Comparison: IcoSema vs Insulin Icodec; Test type: Superiority — Change in HbA1c from baseline to week 52 is analysed using an analysis of covariance (ANCOVA) model with region and randomised treatment as fixed factors and baseline HbA1c as covariate. Missing HbA1c values at week 52 are imputed by using multiple imputation. Each imputed dataset is analysed separately and estimates are combined using Rubin's rules; p < 0.0001, ANCOVA; Treatment difference = -0.66, 95% CI 2-sided [-0.76 to -0.57]

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) to week 52 in body weight is presented. The outcome measure was evaluated based on the data from in study period, where all data from randomisation until last date of any of the following: 1) last direct participant-site contact; 2) participants who withdrew their informed consent; 3) last participant-investigator contact as defined by the investigator for participants who lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death of participants who died before any of the above.
Time Frame: Baseline (Week 0), Week 52
Population: FAS included all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 606 | 610
Kilogram (Kg) | -3.71 (4.87) | 1.96 (4.76)

3. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Less Than 3.0 Millimoles Per Litre [mmol/L] (54 Milligram Per Decilitre [mg/dL]), Confirmed by Blood Glucose [BG] Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Hypoglycaemic episodes were classified according to the American Diabetes Association/ International Hypoglycaemia Study Group, where glycemic criteria for level 2 was less than (<) 3.0 mmol/L (54 mg/dL) and level 3 had no specific glucose threshold. The outcome measure was evaluated based on data from on treatment period, where all data from date of first dose of randomised treatment as recorded on the electronic case report form (eCRF) until the first date of any of the following: 1) last follow-up visit ; 2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after the end of the dosing interval for both treatment arms); 3) end-date for the in-study data points sets.
Time Frame: From baseline week 0 to week 57
Population: Safety analysis set (SAS) included all randomised participants who are exposed to randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 644 | 644
Episodes | 91 | 424

4. Secondary Outcome: Percentage of Time in Range 3.9-10.0 mmol/L (70-180 mg/dL) Using Continuous Glucose Monitoring (CGM) System, Dexcom G6
Description: Time in range was defined as 100 times the number of recorded measurements in glycemic range 3.9-10.0 mmol/L (70-180 mg/dL), both inclusive, divided by the total number of recorded measurements. The outcome measure was evaluated based on the data from in study period: Data from randomisation until last date of any of the following: 1) the last direct participant-site contact; 2) withdrawal for participants who withdraw their informed consent; 3) the last participant-investigator contact as defined by the investigator for participants who are lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death for participants who die before any of the above.
Time Frame: From week 48 to week 52
Population: FAS included all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 481 | 488
Percentage of time | 75.9 (16.1) | 61.9 (18.1)

5. Secondary Outcome: Percentage of Time Spent < 3.0 mmol/L (54 mg/dL) Using Continuous Glucose Monitoring (CGM) System, Dexcom G6
Description: Time spent below threshold was defined as 100 times the number of recorded measurements below the threshold, divided by the total number of recorded measurements. The outcome measure was evaluated based on the data from in study period: Data from randomisation until last date of any of the following: 1) the last direct participant-site contact; 2) withdrawal for participants who withdraw their informed consent; 3) the last participant-investigator contact as defined by the investigator for participants who are lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death for participants who die before any of the above.
Time Frame: From week 48 to week 52
Population: FAS included all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 481 | 488
Percentage of time | 0.27 (0.55) | 0.33 (0.82)

6. Secondary Outcome: Percentage of Time Spent > 10.0 mmol/L (180 mg/dL) Using Continuous Glucose Monitoring (CGM) System, Dexcom G6
Description: Time spent above threshold is defined as 100 times the number of recorded measurements above the threshold, divided by the total number of recorded measurements. The outcome measure was evaluated based on the data from in study period: Data from randomisation until last date of any of the following: 1) the last direct participant-site contact; 2) withdrawal for participants who withdraw their informed consent; 3) the last participant-investigator contact as defined by the investigator for participants who are lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death for participants who die before any of the above.
Time Frame: From week 48 to week 52
Population: FAS included all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 481 | 488
Percentage of time | 23.2 (16.3) | 36.7 (18.7)

7. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline (week 0) to week 52 is presented. The outcome measure was evaluated based on the data from in study period: Data from randomisation until last date of any of the following: 1) the last direct participant-site contact; 2) withdrawal for participants who withdraw their informed consent; 3) the last participant-investigator contact as defined by the investigator for participants who are lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death for participants who die before any of the above.
Time Frame: Baseline (Week 0), Week 52
Population: FAS included all randomised participants. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 552 | 572
Millimoles per litre (mmol/L) | -1.90 (3.01) | -1.65 (2.96)

8. Secondary Outcome: Weekly Basal Insulin Dose
Description: Estimated mean average weekly basal insulin dose from week 50 to week 52 of treatment is presented. The outcome measure was evaluated based on data from on treatment period, where all data from date of first dose of randomised treatment as recorded on the electronic case report form (eCRF) until the first date of any of the following: 1) last follow-up visit (V56); 2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after the end of the dosing interval for both treatment arms); 3) end-date for the in-study data points sets.
Time Frame: From week 50 to week 52
Population: SAS included all randomised participants who are exposed to randomised treatment. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Units of insulin
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 575 | 596
Units of insulin | 170.6 (83.3) | 366.5 (225.5)

9. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter)
Description: Hypoglycaemic episodes were classified according to the American Diabetes Association/ International Hypoglycaemia Study Group, where glycemic criteria for level 2 was less than (<) 3.0 mmol/L (54 mg/dL). The outcome measure was evaluated based on data from on treatment period, where all data from date of first dose of randomised treatment as recorded on the electronic case report form (eCRF) until the first date of any of the following: 1) last follow-up visit ; 2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after the end of the dosing interval for both treatment arms); 3) end-date for the in-study data points sets.
Time Frame: From baseline week 0 to week 57
Population: SAS included all randomised participants who are exposed to randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 644 | 644
Episodes | 90 | 419

10. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Hypoglycaemic episodes were classified according to the American Diabetes Association/ International Hypoglycaemia Study Group, where glycemic criteria for level 3 had no specific glucose threshold. The outcome measure was evaluated based on data from on treatment period, where all data from date of first dose of randomised treatment as recorded on the electronic case report form (eCRF) until the first date of any of the following: 1) last follow-up visit; 2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after the end of the dosing interval for both treatment arms); 3) end-date for the in-study data points sets.
Time Frame: From baseline week 0 to week 57
Population: SAS included all randomised participants who are exposed to randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | IcoSema | Insulin Icodec
Number analyzed (Participants) | 644 | 644
Episodes | 1 | 5

ADVERSE EVENTS:
Time Frame: Week 0 to week 57
Description: Presented AEs are TEAEs, defined as event with onset during on treatment period where all data from date of first dose of randomised treatment as recorded on electronic case report form until first date of any of the below: last follow up visit; last date on random-ised treatment +6 weeks (corresponding to 5 weeks after end of dosing interval for both arms); end-date for in-study data points. AEs were evaluated using SAS. All-Cause Mortality was assessed for all participants enrolled in study.
Groups:
- Icodec: Participants received once-weekly subcutaneous injections of 700 U/mL of insulin icodec for 52 weeks.
Arm/Group | Icodec | IcoSema
All-Cause Mortality (participants affected / at risk) | 3/645 | 2/646
Serious Adverse Events (participants affected / at risk) | 69/644 | 59/644
Other Adverse Events (participants affected / at risk) | 258/644 | 354/644
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icodec (N=644) | IcoSema (N=644)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (4) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Degenerative aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Terminal ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icodec (N=644) | IcoSema (N=644)
COVID-19 (Infections and infestations) | 61 (62) | 67 (68)
Constipation (Gastrointestinal disorders) | 8 (8) | 39 (55)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 38 (48)
Diabetic retinopathy (Eye disorders) | 35 (41) | 41 (46)
Diarrhoea (Gastrointestinal disorders) | 46 (65) | 102 (187)
Dizziness (Nervous system disorders) | 19 (27) | 37 (41)
Dyspepsia (Gastrointestinal disorders) | 10 (11) | 44 (64)
Headache (Nervous system disorders) | 20 (26) | 33 (58)
Nasopharyngitis (Infections and infestations) | 51 (62) | 38 (50)
Nausea (Gastrointestinal disorders) | 24 (29) | 153 (348)
Upper respiratory tract infection (Infections and infestations) | 69 (84) | 54 (64)
Vomiting (Gastrointestinal disorders) | 17 (19) | 68 (118)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT05352815/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT05352815/SAP_001.pdf